CLINICAL TRIAL: NCT04307888
Title: Spanish Percutaneous Aortic INtervention REGISTRY (SPAIN REGISTRY)
Acronym: SPAIN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sociedad Espanola de Angiologia y Cirugia Vascular (Network)
Responsible Party: Sponsor
Other Study IDs: RIV-2019-01
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Aorta Aneurysm; Aorta Dissection; Aorta Stenosis; Aortic Coarctation; Aortic Rupture; Aortic Valve Disease; Aortic Valve Stenosis
Keywords: Percutaneous access
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection; Aortic Valve Stenosis; Aortic Coarctation; Aortic Rupture; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study group: Patients undergoing Percutaneous Endovascular Aneurysm Repair (PEVAR), Percutaneous Endovascular Thoracic Aneurysm Repair (PTEVAR) or Transcatheter Aortic Valve Implantation (TAVI) in who percutaneous access closure device is used for implanting devices at aorta level.
  Interventions: Device: Perclose Proglide (Abbott)

INTERVENTIONS:
Device: Perclose Proglide (Abbott) — Common Femoral Artery percutaneous access closure by means of Perclose Proglide device

SUMMARY:
Multicentre prospective registry including consecutive patients undergoing Percutaneous Endovascular Aneurysm Repair (PEVAR), Percutaneous Endovascular Thoracic Aneurysm Repair (PTEVAR) or Transcatheter Aortic Valve Implantation (TAVI) in which variables related to the percutaneous access closure for implanting devices at aorta level will be collected and analyzed.

The follow-up period will be 30 days after the procedure. The duration of the recruitment period will be one year. All data will be collected telematically and incorporated into a database for subsequent statistical analysis.

There will be 2 points for data interim analysis at 6 and 12 months after initiation of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old
* Signed informed consent
* Endovascular procedures on the aorta to any level, performed by percutaneous access and requiring the use of devices ≥ 10F
* Femoral Access suitable for percutaneous treatment in the opinion of the surgeon

Exclusion Criteria:

* Need for surgical repair of the femoral artery (stenosis aneurysmal)
* Initial indication of percutaneous closure with another device different from the Perclose Proglide
* Active infection of the puncture site
* Condition that prevents complete the 30 days follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Percutaneous Endovascular Aneurysm Repair (PEVAR), Percutaneous Endovascular Thoracic Aneurysm Repair (PTEVAR) or Transcatheter Aortic Valve Implantation (TAVI) in who percutaneous access closure device is used for implanting devices at aorta level.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Rate of closure-procedure technical success as assessed by absence of femoral pseudoaneurysm or arterial occlusion | 30 days
  Rate of cases that are reported with a femoral pseudoaneurysm in the site of arterial access or common femoral artery occlusion related to the closure procedure.
Quality of Life assesed by EuroQol-5 Dimensions (EQ-5D) Questionnaire | 30 days
  Estimated Impact of the procedure on the Quality of Life measured by EQ-5D Questionnaire on 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The study participants self-rate their level of severity for each dimension.
  Rated level can be coded as 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Incidence of Procedure-Emergent Adverse Events related to Frailty as assessed by the Modified Frailty Index (mFI-11) | 30 days
  Incidence of any postoperative adverse event or mortality related to the frailty assessed by the modified frailty index (mFI-11), an 11-factor score predictive of increased risk for postoperative morbidity and mortality in patients undergoing elective and emergent surgery that scores the frailty between 1 to 11, being the 11 the most frailty status.

SECONDARY OUTCOMES:
Time of closure procedure hemostasis in seconds | 1 hour
  Duration in seconds of the arterial closure procedure until complete hemostasis
Hospital Stay assessed in days | 30 days
  Duration in days until hospital discharge
Post-operative Pain assessed by the Visual Analog Scale for Pain | 30 days
  Evaluation of the discomfort or pain after the procedure determined at the end of the procedure with the Visual Analog Scale for Pain, which is a psychometric measuring instrument designed to assess the pain intensity experienced by each patient individually.
  The analogous visual scale used for this study measures from 0-10 the intensity of the pain with a series of "faces" that show the intensity in the pain experimentation with categories like "No pain" approximately 0-1, mild, annoying in number 2, nagging in number 4, distressing in number 6, intense in number 8 and worst possible in number 10.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Hernandez Carbonell, MD, Study Director — Hospital Quiron Salud Marbella; Francisco J Medina, MD, Study Director — Hospital Universitario Burgos; Ignacio Agundez-Gomez, MD, Study Director — Hospital Universitario Burgos

IPD SHARING:
Plan to Share IPD: Undecided